CLINICAL TRIAL: NCT00525369
Title: IL 6 Measurement Using a New Densitometric Bedside (POC) Test
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Other Study IDs: STU-IL-6-1
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-09

CONDITIONS: Sepsis, Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
In a equivalence analysis, we determined whether IL-6 can be assessed using a new densitometric point-of-care (POC) assay (turn-around -time: 20 minutes).IL-6 measurements were compared to test results obtained with conventional ELISA analysis

DETAILED DESCRIPTION:
In an equivalence analysis, we determined whether IL-6 can be assessed using a new densitometric point-of-care (POC) assay (turn-around -time: 20 minutes) that allows IL-6 measurements at the bedside. We then compared the respective test results to those obtained with conventional ELISA analysis

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Written informed consent

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Georg Schlosser, MD, Principal Investigator — Charite University, Berlin, Germany; Joerg C Schefold, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite University Medicine Berlin, Berlin, State of Berlin, Germany